CLINICAL TRIAL: NCT02278081
Title: The Relationship Between Gastroesophageal Reflux and Pediatric Rhinitis: Significance of Pale/Blue Colored Turbinate. A Randomized Controlled Trial
Brief Title: The Relationship Between Gastroesophageal Reflux and Pediatric Rhinitis: Significance of Pale/Blue Colored Turbinate
Acronym: Pale Turbinate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, John Manoukian, Associate Professor, Faculty of Medicine, McGill University, Department of Otolaryngology-Head and Neck Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4225
Record Dates: First submitted 2014-10-21; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Rhinitis; Nasal Obstruction; GERD
Keywords: Rhinitis (nasal obstruction) and GERD
MeSH Terms: conditions — Rhinitis; Nasal Obstruction; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Experimental): The treatment group will receive 30 mg lansoprazole (prevacid) one capsule per day for three months and mometasone furonate (nasonex) one puff in each nostril per day for three months.
  Interventions: Drug: lansoprazole
- placebo group (Placebo Comparator): The placebo group will receive one capsule per day of prevacid placebo for three months and mometasone furonate (nasonex) one puff in each nostril per day for three months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lansoprazole — the lansoprazole will be taken orally.
  Arms: treatment group
Drug: placebo — the lansoprazole placebo will be taken orally.
  Arms: placebo group

SUMMARY:
Gastroesophageal(GERD) reflux disease is a very common problem among pediatric population and has be proved to contribute in numerous otolaryngological manifestations. Trails of empirical treatment of antireflux medications is often used as a diagnostic test. However, the investigators believe GERD can cause rhinitis and nasal obstruction. Nasonex is considered as first line treatment for nasal obstruction. Hence, the proposed study aims to define the relationship between GERD and rhinitis using randomize control trial where one group of patients will receive nasonex and placebo, while the other group will receive nasonex and antireflux medications.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial in which children with nasal obstruction will be randomized to receive either antireflux medication lansoprazole (prevacid) and mometasone furonate (nasonex) or only nasonex and placebo. The diagnosis of nasal obstruction will be made by history and physical examination.

The study will take place at Montreal children's hospital. After the patients or parents of the patients agree for their children to take part in the study and sign a consent/assent form, baseline information will be collected and the patients will asked to fill out three questionnaires for GERD symptoms and nasal symptom. After that eligible patients will undergo sinus x-ray, nasal endoscopy and allergy skin test (these test are routine performed for all patients with symptoms of nasal obstruction). Then the patients will further be sub-divided into two groups based on the allergic skin prick test (SPT); allergy positive and allergy negative group. In each group patients will randomly allocated to one of the two study arms; group A will receive lansoprazole (prevacid) and mometasone furonate (nasonex) and the other group will receive nasonex and placebo. The lansoprazole/placebo will be discontinued after 3 months and the patients will undergo nasal endoscopy and will be asked to fill out the three questionnaires again to assess the improvement. The patients will be follow for another 3 months, the patients will again undergo nasal endoscopy and will asked to fill out the three questionnaires to assess the improvement and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* 7 (seven) to 17 (seventeen) years of age.
* Nasal obstruction as main complaint.

Exclusion Criteria:

* Structural cause of nasal obstruction (deviated nasal septum, adenoid hypertrophy, nasal polyps, nasal tumors)
* Received antireflux medication during the last three months.
* Acute sinusitis

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
improvement of the nasal signs and symptoms. | three months
  after three months of treatment the patient symptoms will be evaluated using subjective questionnaires and nasal endoscopic exam .

REFERENCES:
- [Background] Vandenplas Y, Rudolph CD, Di Lorenzo C, Hassall E, Liptak G, Mazur L, Sondheimer J, Staiano A, Thomson M, Veereman-Wauters G, Wenzl TG, North American Society for Pediatric Gastroenterology Hepatology and Nutrition, European Society for Pediatric Gastroenterology Hepatology and Nutrition. Pediatric gastroesophageal reflux clinical practice guidelines: joint recommendations of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition (NASPGHAN) and the European Society for Pediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN). J Pediatr Gastroenterol Nutr. 2009 Oct;49(4):498-547. doi: 10.1097/MPG.0b013e3181b7f563. PMID 19745761
- [Background] Zalzal GH, Tran LP. Pediatric gastroesophageal reflux and laryngopharyngeal reflux. Otolaryngol Clin North Am. 2000 Feb;33(1):151-61. doi: 10.1016/s0030-6665(05)70212-7. PMID 10637349
- [Background] Ali Mel-S. Laryngopharyngeal reflux: diagnosis and treatment of a controversial disease. Curr Opin Allergy Clin Immunol. 2008 Feb;8(1):28-33. doi: 10.1097/ACI.0b013e3282f3f44f. PMID 18188014
- [Background] Karkos PD, Leong SC, Apostolidou MT, Apostolidis T. Laryngeal manifestations and pediatric laryngopharyngeal reflux. Am J Otolaryngol. 2006 May-Jun;27(3):200-3. doi: 10.1016/j.amjoto.2005.09.004. PMID 16647985
- [Background] Al-Saab F, Manoukian JJ, Al-Sabah B, Almot S, Nguyen LH, Tewfik TL, Daniel SJ, Schloss MD, Hamid QA. Linking laryngopharyngeal reflux to otitis media with effusion: pepsinogen study of adenoid tissue and middle ear fluid. J Otolaryngol Head Neck Surg. 2008 Aug;37(4):565-71. PMID 19128594
- [Background] Contencin P, Maurage C, Ployet MJ, Seid AB, Sinaasappel M. Gastroesophageal reflux and ENT disorders in childhood. Int J Pediatr Otorhinolaryngol. 1995 Jun;32 Suppl:S135-44. doi: 10.1016/0165-5876(94)01157-s. PMID 7665283
- [Background] El-Serag HB, Gilger M, Kuebeler M, Rabeneck L. Extraesophageal associations of gastroesophageal reflux disease in children without neurologic defects. Gastroenterology. 2001 Dec;121(6):1294-9. doi: 10.1053/gast.2001.29545. PMID 11729108
- [Background] Yuksel F, Dogan M, Karatas D, Yuce S, Senturk M, Kulahli I. Gastroesophageal reflux disease in children with chronic otitis media with effusion. J Craniofac Surg. 2013 Mar;24(2):380-3. doi: 10.1097/SCS.0b013e31827feb08. PMID 23524698
- [Background] Nair S, Kumar M, Nair P. Role of GERD in children with otitis media with effusion. Indian J Pediatr. 2012 Oct;79(10):1328-32. doi: 10.1007/s12098-011-0671-y. Epub 2012 Jan 7. PMID 22227976
- [Background] Benninger MS, Ferguson BJ, Hadley JA, Hamilos DL, Jacobs M, Kennedy DW, Lanza DC, Marple BF, Osguthorpe JD, Stankiewicz JA, Anon J, Denneny J, Emanuel I, Levine H. Adult chronic rhinosinusitis: definitions, diagnosis, epidemiology, and pathophysiology. Otolaryngol Head Neck Surg. 2003 Sep;129(3 Suppl):S1-32. doi: 10.1016/s0194-5998(03)01397-4. No abstract available. PMID 12958561
- [Background] Phipps CD, Wood WE, Gibson WS, Cochran WJ. Gastroesophageal reflux contributing to chronic sinus disease in children: a prospective analysis. Arch Otolaryngol Head Neck Surg. 2000 Jul;126(7):831-6. doi: 10.1001/archotol.126.7.831. PMID 10888994
- [Background] Lupa M, DelGaudio JM. Evidence-based practice: reflux in sinusitis. Otolaryngol Clin North Am. 2012 Oct;45(5):983-92. doi: 10.1016/j.otc.2012.06.004. Epub 2012 Aug 9. PMID 22980679
- [Background] Loehrl TA, Smith TL, Darling RJ, Torrico L, Prieto TE, Shaker R, Toohill RJ, Jaradeh SS. Autonomic dysfunction, vasomotor rhinitis, and extraesophageal manifestations of gastroesophageal reflux. Otolaryngol Head Neck Surg. 2002 Apr;126(4):382-7. doi: 10.1067/mhn.2002.123857. PMID 11997777